CLINICAL TRIAL: NCT00469859
Title: A Pilot Study of Lestaurtinib (CEP-701) in Combination With Chemotherapy in Young Patients With Relapsed or Refractory FLT3-mutant Acute Myeloid Leukemia
Brief Title: Lestaurtinib, Cytarabine, and Idarubicin in Treating Younger Patients With Relapsed or Refractory Acute Myeloid Leukemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAML06P1; CDR0000543398 (Other: Clinical Trials.gov); COG-AAML06P1 (Other: Children's Oncology Group)
Record Dates: First submitted 2007-05-03; First posted 2007-05-07 (Estimated); Results first posted 2013-12-20 (Estimated); Last update posted 2017-03-15 (Actual); Status verified 2017-02

CONDITIONS: Leukemia
Keywords: recurrent childhood acute myeloid leukemia; adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); recurrent adult acute myeloid leukemia; secondary acute myeloid leukemia
MeSH Terms: conditions — Leukemia; Congenital Abnormalities; Leukemia, Myeloid, Acute | interventions — Cytarabine; Idarubicin; lestaurtinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Lestaurtinib dose 50 mg/m2 (Experimental): DOSE-FINDING PHASE:
  COURSE 1: Patients receive cytarabine IV over 2 hours twice daily on days 1-4, idarubicin IV over 15 minutes on days 2-4, and oral lestaurtinib twice daily on days 5-28. Patients achieving complete or partial response proceed to course 2. Cohorts of 6 patients receive escalating doses of lestaurtinib until a TBAD is determined. The TBAD is defined as the dose at which no more than 2 of 6 patients experience DLT and biologic activity is confirmed by PIA assay.
  COURSE 2: Patients receive high-dose cytarabine IV over 3 hours twice daily on days 1-4 and oral lestaurtinib (at the dose determined in course 1) twice daily on days 5-28. Patients achieving complete or partial response proceed to continuation therapy.
  CONTINUATION THERAPY: Patients receive oral lestaurtinib twice daily on days 1-28. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Continued (see detailed description)
  Interventions: Drug: cytarabine; Drug: idarubicin; Drug: lestaurtinib
- Group 2 (Lestaurtinib: Dose 62.5 mg/m2 (Experimental): DOSE-FINDING PHASE:
  COURSE 1: Patients receive cytarabine IV over 2 hours twice daily on days 1-4, idarubicin IV over 15 minutes on days 2-4, and oral lestaurtinib twice daily on days 5-28. Patients achieving complete or partial response proceed to course 2. Cohorts of 6 patients receive escalating doses of lestaurtinib until a TBAD is determined. The TBAD is defined as the dose at which no more than 2 of 6 patients experience DLT and biologic activity is confirmed by PIA assay.
  COURSE 2: Patients receive high-dose cytarabine IV over 3 hours twice daily on days 1-4 and oral lestaurtinib (at the dose determined in course 1) twice daily on days 5-28. Patients achieving complete or partial response proceed to continuation therapy.
  CONTINUATION THERAPY: Patients receive oral lestaurtinib twice daily on days 1-28. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Continued (see detailed description)
  Interventions: Drug: cytarabine; Drug: idarubicin; Drug: lestaurtinib

INTERVENTIONS:
Drug: cytarabine — given IV
  Other Names: Cytosine arabinoside; Ara-C; Cytosar; NSC #063878
Drug: idarubicin — Given IV
  Other Names: Idarubicin HCl; 4-Demethoxydaunorubicin; 4-DMD; DMDR; IdamycinPFS
Drug: lestaurtinib — Given orally
  Other Names: benzodiazocin-1-one; IND#76431

SUMMARY:
RATIONALE: Lestaurtinib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as cytarabine and idarubicin, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving lestaurtinib together with cytarabine and idarubicin may kill more cancer cells.

PURPOSE: This phase I/II trial is studying the side effects and best dose of lestaurtinib when given together with cytarabine and idarubicin and to see how well they work in treating younger patients with relapsed or refractory acute myeloid leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine a safe, tolerable, and biologically active dose of lestaurtinib in combination with chemotherapy comprising cytarabine and idarubicin in younger patients with relapsed or refractory FLT3-mutant acute myeloid leukemia.

Secondary

* Determine the overall response rate in patients treated with this regimen.
* Optimize dosing of lestaurtinib based primarily on biologic activity rather than toxicity.
* Correlate the clinical response to this regimen with the ability to achieve adequate FLT3 plasma inhibitory activity levels and the in vitro sensitivity of pretreatment leukemic cells to lestaurtinib in these patients.
* Determine the mechanisms of resistance to lestaurtinib in these patients.
* Assess the feasibility of using rapid central determination of FLT3 mutation status at study entry to determine induction therapy in future upfront protocols.

OUTLINE: This is a multicenter, dose-finding study of lestaurtinib followed by an efficacy study.

* Dose-finding phase:

  * Course 1: Patients receive cytarabine IV over 2 hours twice daily on days 1-4, idarubicin IV over 15 minutes on days 2-4, and oral lestaurtinib twice daily on days 5-28. Patients achieving complete or partial response proceed to course 2.

Cohorts of 6 patients receive escalating doses of lestaurtinib until a tolerable and biologically active dose (TBAD) is determined. The TBAD is defined as the dose at which no more than 2 of 6 patients experience DLT and biologic activity is confirmed by plasma inhibitory activity (PIA) assay.

* Course 2: Patients receive high-dose cytarabine IV over 3 hours twice daily on days 1-4 and oral lestaurtinib (at the dose determined in course 1) twice daily on days 5-28. Patients achieving complete or partial response proceed to continuation therapy.
* Continuation therapy: Patients receive oral lestaurtinib twice daily on days 1-28. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

  * Efficacy phase: Once the TBAD is determined, subsequent patients receive treatment as in course 1 and 2 with lestaurtinib at the TBAD. Patients may also receive continuation therapy as in the dose-finding phase.

Blood samples are collected periodically during study treatment for pharmacokinetic and PIA assays.

After completion of study treatment, patients are followed periodically for up to 5 years.

PROJECTED ACCRUAL: A total of 37 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of acute myeloid leukemia (AML) according to FAB classification

  * At least 5% blasts in the bone marrow, with or without extramedullary disease
* In first relapse after induction therapy OR refractory to induction therapy with ≤ 1 attempt at remission induction

  * Patients who are in a first relapse > 1 year from their initial diagnosis of AML are excluded from the dose-finding phase of the study, but are eligible for the efficacy phase
  * First relapse after hematopoietic stem cell transplantation (HSCT) allowed provided patient has no evidence of active graft-versus-host disease (GVHD) and is at least 4 months posttransplantation
* Positive for a FLT3 activating mutation (internal tandem duplication or kinase domain point mutation) using standard polymerase chain reaction-based procedures at any time in the course of illness
* Treatment-related AML allowed

PATIENT CHARACTERISTICS:

* Karnofsky performance status (PS) 50-100% (> 16 years of age) OR Lansky PS 50-100% (≤ 16 years of age)
* Creatinine clearance or radioisotope glomerular filtration rate ≥ 70 mL/min OR serum creatinine based on age and gender as follows:

  * Creatinine no greater than 0.4 mg/dL (1 month to < 6 months of age)
  * Creatinine no greater than 0.5 mg/dL (6 months to < 1 year of age)
  * Creatinine no greater than 0.6 mg/dL (1 year to < 2 years of age)
  * Creatinine no greater than 0.8 mg/dL (2 years to < 6 years of age)
  * Creatinine no greater than 1 mg/dL (6 years to < 10 years of age)
  * Creatinine no greater than 1.2 mg/dL (10 years to < 13 years of age)
  * Creatinine no greater than 1.4 mg/dL (females) or 1.5 mg/dL (males) (13 years to < 16 years of age)
  * Creatinine no greater than 1.4 mg/dL (females) or 1.7 mg/dL (males) (16 years of age and over)
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* ALT < 5 times ULN (unless it is related to leukemic involvement)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Shortening fraction ≥ 27% by echocardiogram OR ejection fraction ≥ 50% by radionuclide angiogram

PRIOR CONCURRENT THERAPY:

* Recovered from all prior therapy
* No prior cumulative anthracycline doses exceeding 450 mg/m^2 daunorubicin equivalents

  * Patients who relapse after receiving treatment on protocol COG-AAML03P1 or COG-AAML0531 (300 mg/m^2 of daunorubicin hydrochloride and 48 mg/m^2 of mitoxantrone hydrochloride) allowed provided they have not received any additional anthracyclines
* At least 14 days since prior cytotoxic therapy

  * Hydroxyurea allowed to decrease the WBC prior to starting protocol treatment
  * No concurrent hydroxyurea
* At least 7 days since prior biologic agents
* At least 14 days since prior monoclonal antibody therapy
* Radiotherapy to chloromas allowed

  * Irradiated lesion may not be used to assess tumor response
* No other concurrent chemotherapy, investigational therapy, immunomodulating agents, or steroids

  * Steroids used as an antiemetic allowed
  * Prophylactic intrathecal cytarabine allowed
* No concurrent CYP3A4,5 inhibitors, including any of the following:

  * Azole antifungals (e.g., fluconazole or voriconazole)
  * Cyclosporine
  * Erythromycin
  * Clarithromycin
  * Troleandomycin
  * HIV protease inhibitors
  * Nefazodone
* No concurrent CYP3A4,5 inducers, including any of the following:

  * Carbamazepine
  * Dexamethasone
  * Rifampin
  * Phenobarbital
  * Phenytoin
  * Hypericum perforatum (St. John's wort)

Ages: 1 Year to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 14 (Actual)
Dates: Start 2007-06; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick A. Brown, MD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins; Donald Small, MD, PhD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (21):
- United States (21):
  - Lurleen Wallace Comprehensive Cancer at University of Alabama - Birmingham, Birmingham, Alabama
  - Children's Hospital of Orange County, Orange, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Children's Memorial Hospital - Chicago, Chicago, Illinois
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - C.S. Mott Children's Hospital at University of Michigan Medical Center, Ann Arbor, Michigan
  - Masonic Cancer Center at University of Minnesota, Minneapolis, Minnesota
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - Herbert Irving Comprehensive Cancer Center at Columbia University Medical Center, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Knight Cancer Institute at Oregon Health and Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Simmons Comprehensive Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - Baylor University Medical Center - Houston, Houston, Texas
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1 (Lestaurtinib Dose 50 mg/m2): COURSE 1: Cytarabine IV over 2 hours twice daily days 1-4, idarubicin IV over 15 minutes days 2-4, and oral lestaurtinib twice daily days 5-28. Patients achieving complete or partial response proceed to course 2. Cohorts of 6 patients receive escalating doses of lestaurtinib until a safe, tolerable and biologically active dose (TBAD) is determined. The TBAD is defined as the dose at which no more than 2 of 6 patients experience DLT and biologic activity is confirmed by PIA assay.
  COURSE 2: Patients receive high-dose cytarabine IV over 3 hours twice daily days 1-4 and oral lestaurtinib (at the dose determined in course 1) twice daily days 5-28. Patients achieving complete or partial response proceed to continuation therapy.
  CONTINUATION THERAPY: Patients receive oral lestaurtinib twice daily days 1-28. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Continued (see detailed description)
- Group 2 (Lestaurtinib: Dose 62.5 mg/m2): COURSE 1: Cytarabine IV over 2 hours twice daily days 1-4, idarubicin IV over 15 minutes days 2-4, and oral lestaurtinib twice daily days 5-28. Patients achieving complete or partial response proceed to course 2. Cohorts of 6 patients receive escalating doses of lestaurtinib until a safe, tolerable and biologically active dose (TBAD) is determined. The TBAD is defined as the dose at which no more than 2 of 6 patients experience DLT and biologic activity is confirmed by PIA assay.
  COURSE 2: Patients receive high-dose cytarabine IV over 3 hours twice daily days 1-4 and oral lestaurtinib (at the dose determined in course 1) twice daily days 5-28. Patients achieving complete or partial response proceed to continuation therapy.
  CONTINUATION THERAPY: Patients receive oral lestaurtinib twice daily on days 1-28. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Continued (see detailed description)
  cytarabine
Period: Overall Study
Arm/Group | Group 1 (Lestaurtinib Dose 50 mg/m2) | Group 2 (Lestaurtinib: Dose 62.5 mg/m2)
Started | 6 | 8
Completed | 6 | 6
Not Completed | 0 | 2
Not completed — Inevaluable | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Group 1 (Lestaurtinib Dose 50 mg/m2; Group 2 (Lestaurtinib: Dose 62.5 mg/m2: COURSE 1: Patients receive cytarabine IV over 2 hours twice daily on days 1-4, idarubicin IV over 15 minutes on days 2-4, and oral lestaurtinib twice daily on days 5-28. Patients achieving complete or partial response proceed to course 2. Cohorts of 6 patients receive escalating doses of lestaurtinib until a TBAD is determined. The TBAD is defined as the dose at which no more than 2 of 6 patients experience DLT and biologic activity is confirmed by PIA assay.
  COURSE 2: Patients receive high-dose cytarabine IV over 3 hours twice daily on days 1-4 and oral lestaurtinib (at the dose determined in course 1) twice daily on days 5-28. Patients achieving complete or partial response proceed to continuation therapy.
  CONTINUATION THERAPY: Patients receive oral lestaurtinib twice daily on days 1-28. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Continued (see detailed description)
- Total: Total of all reporting groups
Arm/Group | Group 1 (Lestaurtinib Dose 50 mg/m2 | Group 2 (Lestaurtinib: Dose 62.5 mg/m2 | Total
Number analyzed (Participants) | 6 | 8 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6 | 8 | 14
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 2 | 6 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 4 | 8 | 12
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 4 | 5 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 8 | 14

OUTCOME MEASURES:

1. Primary Outcome: Dose-limiting Toxicity
Description: Number of patients with dose-limiting toxicity (DLT)
Time Frame: 28 days
Measure: Number; unit: participants
Arm/Group | Group 1 (Lestaurtinib Dose 50 mg/m2 | Group 2 (Lestaurtinib: Dose 62.5 mg/m2
Number analyzed (Participants) | 6 | 6
participants | 0 | 0

2. Primary Outcome: >80% Inhibition of FLT3 Phosphorylation in a Majority of Post-treatment Trough Time Points
Description: FLT3 inhibition is determined in patients receiving lestaurtinib by measuring FLT3 plasma inhibitory activity (PIA). For PIA predictive modeling, a random effects linear regression model will be used to describe the relationship between PIA and Pharmacokinetic (PK) levels for each of the 5 trough plasma samples collected for each patient
Time Frame: Course 1 day 7, day 14, day 21, and day 28.
Measure: Number; unit: participants
Arm/Group | Group 1 (Lestaurtinib Dose 50 mg/m2 | Group 2 (Lestaurtinib: Dose 62.5 mg/m2
Number analyzed (Participants) | 6 | 6
participants | 5 | 5

ADVERSE EVENTS:
Arm/Group | Group 1 (Lestaurtinib Dose 50 mg/m2 | Group 2 (Lestaurtinib: Dose 62.5 mg/m2
Serious Adverse Events (participants affected / at risk) | 2/6 | 6/8
Other Adverse Events (participants affected / at risk) | 6/6 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (Lestaurtinib Dose 50 mg/m2 (N=6) | Group 2 (Lestaurtinib: Dose 62.5 mg/m2 (N=8)
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Acidosis (Metabolism and nutrition disorders) | 0 | 1
Activated partial thromboplastin time prolonged (Investigations) | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1
Alkalosis (Metabolism and nutrition disorders) | 0 | 1
Anemia (Blood and lymphatic system disorders) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 3
Anxiety (Psychiatric disorders) | 0 | 1
Appendicitis perforated (Infections and infestations) | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Cardiac disorders - Other (Cardiac disorders) | 0 | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 1 | 4
Hypotension (Vascular disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Infections and infestations - Other (Infections and infestations) | 1 | 4
Intracranial hemorrhage (Nervous system disorders) | 0 | 1
Left ventricular systolic dysfunction (Cardiac disorders) | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 1
Mucositis oral (Gastrointestinal disorders) | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 1
Platelet count decreased (Investigations) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1
Seizure (Nervous system disorders) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 1
Typhlitis (Gastrointestinal disorders) | 0 | 1
Weight gain (Investigations) | 0 | 1
White blood cell decreased (Investigations) | 0 | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (Lestaurtinib Dose 50 mg/m2 (N=6) | Group 2 (Lestaurtinib: Dose 62.5 mg/m2 (N=8)
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Alanine aminotransferase increased (Investigations) | 2 | 1
Anemia (Blood and lymphatic system disorders) | 3 | 6
Anorexia (Metabolism and nutrition disorders) | 1 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 3
Fever (General disorders) | 0 | 1
Hemorrhoids (Gastrointestinal disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 2
Hypokalemia (Metabolism and nutrition disorders) | 1 | 2
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Infections and infestations - Other (Infections and infestations) | 1 | 2
Lipase increased (Investigations) | 0 | 1
Lymphocyte count decreased (Investigations) | 1 | 5
Nausea (Gastrointestinal disorders) | 1 | 1
Neutrophil count decreased (Investigations) | 4 | 5
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Platelet count decreased (Investigations) | 4 | 6
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 1
Rectal pain (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 1
Uterine hemorrhage (Reproductive system and breast disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1
Weight loss (Investigations) | 0 | 1
White blood cell decreased (Investigations) | 4 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Must obtain prior Sponsor approval.